CLINICAL TRIAL: NCT05528731
Title: Perception of Female Hormonal Contraception by the Main Prescribers
Acronym: CHF
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8637
Record Dates: First submitted 2022-09-02; First posted 2022-09-06 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Female Hormonal Contraception
Keywords: Female Hormonal Contraception

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The recommendations for contraception, after researching contraindications to certain methods, are to offer clear and honest information to allow the patient to make an informed choice, adapted to her lifestyle. The best contraception is the one chosen by the patient. The choice of contraception illustrates the difficulty of assessing the benefit-risk balance in the context of functional and preventive treatment.

Taking into account this imbalance between patient beliefs and medical advice is an essential step in improving the provision of gynecological care.

ELIGIBILITY:
Inclusion criteria:

* Any health care professional in general medicine, gynecology and midwifery
* graduate or in progress
* in practice (any practice modality in metropolitan France)
* agreeing to participate in the survey by completing the questionnaire anonymously, after having read the information and non-objection notice attached to the questionnaire.

Exclusion criteria:

- Any other health profession

Inclusion criteria:

- Any health care professional in general medicine, gynecology and midwifery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any health care professional in general medicine, gynecology and midwifery, graduate or in progress in practice (any practice modality in metropolitan France)
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Study of the perception of risks and management of adverse effects of hormonal contraception among prescribers | 5 months after interviews with prescribers

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Assistance Médicale à la Procréation - CHU de Strasbourg - France, Strasbourg, France